CLINICAL TRIAL: NCT03345602
Title: Evaluation of the Serum S100B Protein Assay in the Management of Mild Head Injury Under Anticoagulation
Brief Title: Serum S100B Protein Assay in Mild Head Injury
Acronym: TCLAS-100B
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 17-091
Record Dates: First submitted 2017-11-03; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Light Head Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum S100B protein assay measurement — serum S100B protein assay measurement within the 3 hours after head trauma

SUMMARY:
Head injuries are a major public health issue, with an estimated annual incidence in Europe of 262 per 100,000 population. Light head injury (SCI), defined by a Glasgow score between 13 and 15, constitutes the majority (71% to 98%) of head injury cases. Despite a generally good prognosis, patients with TCL have a low but real risk of brain damage, whose prevalence is estimated at 5%. Cerebral computed tomography (CT) because of its high sensitivity for the detection of posttraumatic intracranial lesions (LIC), is currently considered the gold standard for the diagnosis of these lesions in patients considered at risk after clinical evaluation. The number of cTCTs performed is high with no lesion in more than 90% of cases. The S100B protein, a marker of brain tissue damage, is reported to reliably exclude the presence of brain lesions in adults as well as antiaggregants. These numerous studies show that its serum assay in combination with the clinical decision algorithms allows, thanks to a sensitivity close to 100% for brain lesions, to reduce the number of CTMc currently prescribed by approximately 30%, and therefore to decrease unnecessary exposure to radiation. Although there is no study on the subject, a gain on the duration of care in emergencies can be expected as well as a reduction on the cost of care by a dosage price three times less higher than the TDMc. Expert opinion for the use of this assay in the management of moderate-risk TCL at threshold ≤ 0.10 μg / L in 3h post-TC to ensure sensitivity of 100%, was published in 2014 in the Annales Françaises de Médecine d'Urgence.

The use of anticoagulants has continued to increase in recent years. In 2013, it is estimated that 3.12 million patients received at least one anticoagulant in France. Currently, the international and French recommendations indicate the achievement of cTCT in anticoagulated TCL because it is an independent risk factor for cerebral injury and is therefore considered to be a high risk TCL. LIC. The hypothesis of this study is that the S100B protein assay could also exclude the presence of brain lesion after TCL under anticoagulation in adults

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Emergency department patient with mild head trauma (13 ≤ Glasgow score ≤ 15)
* Affiliated to the social security scheme
* Patient having been informed about the study and do not disagree to participate
* Patient on anticoagulant therapy (enteral or parenteral route)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Cranial Trauma having induced a Glasgow <13
  * Presence of a high risk factor to perform a brain scan (formal indication of cTCT): Focused neurological deficit, Glasgow score <15 at 2 hr, suspicion of open skull fracture or embarrassment, all Sign of fracture of the base of the skull (hemotympanum, bilateral periorbital ecchymosis), otorrhea or rhinorrhea of CSF, convulsion post traumatic.
  * Cranial Trauma time unknown
  * Fuzzy anamnesis
  * Traumatized severe / polytraumatized (victim of a violent trauma, according to the kinetic criteria of Vittel, whatever are the apparent lesions and / or 2 lesions or more of which at least one threatens the vital prognosis)
  * Refusal to participate
  * Refusal to perform a TDMc
  * Congenital or acquired coagulopathy
  * Decision not to carry out a TDMc
  * Active melanoma
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
S100B protein serum concentration | baseline (maximum 3 hours after head trauma)
  The main objective of this study is to evaluate whether a negative serum assay of S100B protein (≤ 0.10 μg / L) within 3 hours after head trauma

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No